CLINICAL TRIAL: NCT06913023
Title: Semaglutide for the Prevention Of Post-Transplant Diabetes Mellitus
Acronym: SPOT-DM
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Sunita Singh, MD, MSc, FRCPC, Principal Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-5093
Record Dates: First submitted 2025-03-17; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Kidney Transplant Recipient
MeSH Terms: interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: This study will use a randomized, double-blind, placebo-controlled clinical trial approach comparing semaglutide to placebo in 50 KTR at risk for PTDM. Adult KTR between 4 and 12 weeks after transplant with an eGFR of at least 30 ml/min/1.73m2 at risk for PTDM will be randomized in a 1:1 fashion to either 24 weeks of semaglutide or 24 weeks of placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Experimental): Patients will be up-titrated as tolerated starting at 3 mg oral semaglutide once daily for 4 weeks, followed by 7 mg oral semaglutide once daily for 4 weeks and then 14 mg oral semaglutide once daily for 16 weeks. Semaglutide can be down-titrated to previously tolerated dose if the current dose is not tolerated by the participant.
  Interventions: Drug: Semaglutide 3 MG [Rybelsus]; Drug: Semaglutide 7 MG [Rybelsus]; Drug: Semaglutide 14 MG [Rybelsus]
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Semaglutide 3 MG [Rybelsus] — Semaglutide 3mg for 4 weeks.
  Arms: Semaglutide
Drug: Semaglutide 7 MG [Rybelsus] — Semaglutide 7mg for 4 weeks.
  Arms: Semaglutide
Drug: Semaglutide 14 MG [Rybelsus] — Semaglutide 14mg for 16 weeks.
  Arms: Semaglutide
Drug: Placebo Oral Tablet — Placebo tablet
  Arms: Placebo

SUMMARY:
The study aims to determine the short-term efficacy, mechanisms and safety of 24 weeks of placebo and semaglutide therapy in 74 KTR at risk of post-transplant diabetes mellitus (PTDM).

DETAILED DESCRIPTION:
A kidney transplant is the best treatment for people living with kidney failure as it allows people to live longer with a better quality of life. However, one in four kidney transplant recipients will develop diabetes after transplant. This is largely due to the medications that must be used to prevent rejection of the transplant. Kidney transplant recipients who get diabetes after transplant are up to three times more likely to have heart disease and die prematurely. To date, there are no treatments to prevent the development of diabetes after kidney transplant. Semaglutide is a drug that is commonly used to treat diabetes and obesity. The investigators believe that semaglutide is a safe and effective drug which can prevent the development of diabetes in kidney transplant recipients. Therefore, the investigators are conducting a study where kidney transplant recipients who are at increased risk of developing diabetes after transplant are randomly assigned to receive either semaglutide or placebo for 24 weeks after their transplant. The study will determine whether semaglutide is effective in decreasing blood sugar levels and the rate of diabetes. The investigators will also study other important markers of health including body weight and cholesterol levels as well as liver, kidney and heart function. Diabetes after transplant is a common problem, and preventing it is extremely important to allowing kidney transplant recipients to live longer and better lives. The results of this study will allow the investigators to determine if semaglutide is a safe and effective option for the prevention of diabetes in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent.
2. Adult (≥18 years) recipients of a living or deceased donor kidney transplant
3. Between 4- and 12-weeks post kidney transplant
4. Stable kidney function defined as an eGFR > 30 ml/min/1.73m2 (CKD-EPI)
5. At risk for PTDM at the time of transplant based on the following criteria:

   1. BMI ≥ 25 kg/m2, or
   2. Fasting plasma glucose 6.1-6.9 mmol/L (impaired fasting glucose), or
   3. 2hr OGTT plasma glucose 7.8-11.0 (impaired glucose tolerance), or
   4. HbA1C 5.5-6.4% (at risk for DM or prediabetes).

Exclusion Criteria:

1. Established diagnosis of type 1 or type 2 DM as per Diabetes Canada (including the need for glucose-lowering therapy for hyperglycemia at the time of screening)
2. Kidney-Pancreas transplant recipient
3. Acute coronary syndrome, transient ischemic attack or stroke within 30 days prior to screening
4. History of pancreatitis
5. Personal or family history of medullary thyroid cancer or MEN2B
6. Women who are pregnant, nursing or plan on becoming pregnant whilst in the trial
7. Use of GLP1RA in the 30 days prior to screening
8. Contraindication to MRI (applicable only to those undergoing the optional MRI assessments)
9. With known or suspected hypersensitivity to semaglutide or related products
10. Patient not able to understand and comply with study requirements, based on Investigator's judgment.
11. Any other clinical condition that, based on Investigator's judgement, would jeopardize patient safety during trial participation or would affect the study outcom
12. History of glucose-galactose malabsorption syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
2-hour OGTT | 24 weeks
  The primary outcome of this study is the change in plasma glucose at 120 minutes following a 75g oral glucose challenge (2-hour OGTT) at 24 weeks. The 2-hour OGTT was selected as the primarily outcome in this study for the following reasons: 1) In selecting a surrogate outcome for PTDM in KTR, there are limitations to HbA1c and fasting glucose in this population; 2) The 2-hour OGTT is the recommended test for the diagnosis of PTDM in KTR and 3) The use of OGTT has been used in other PTDM prevention studies.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 24 weeks
  : The side effects of GLP-1RA have been well described and will be assessed at each study visit. Adverse events include AKI, hypoglycemia, volume depletion, GI intolerance, amputations, pancreatitis, hepatobiliary complications and injection site or allergic reactions, infectious complications (any source), and malignancy. Episodes of biopsy-proven acute rejection (as defined by the Banff criteria), death-censored graft failure (defined as the need for initiation of chronic dialysis or re-transplantation) or death with graft function (defined as death with a functioning allograft) will also be collected. Kidney transplantation assures complete denervation of the transplanted kidney and the renal vasoconstrictive response in the setting of intravascular volume depletion is diminished in KTR. Therefore, frequent monitoring for adverse events has been integrated in our study design, occurring on 10 separate occasions, to capture these adverse events should they occur.
Estimated GFR | 24 weeks
  Calculated by CKD-EPI 2021 equation
Change in fasting blood glucose | 24 weeks
GFR | 24 weeks
  Measured using 24-urine collection for creatinine, standardized per 1.73m2 body surface area. And estimated using CKD-EPI 2021 equation.
Urinary glucose excretion | 24 weeks
  Measured using a 24-hour urine collection for glucose
Change in serum insulin | 24 weeks
Change in HbA1c | 24 weeks
Albuminuria | 24 weeks
  measuring urine albumin excretion from a 24-hour urine collection
Natriuresis | 24 weeks
  Assessed with a 24-hour urine collection for sodium excretion
Percentage of body fat | 24 weeks
  Bioimpedance analysis
Change in fasting lipid profile | 24 weeks
Change in liver enzymes | 24 weeks
  ALT and AST
Change in fibrosis level | 24 weeks
  Transient elastography
Change in steatosis level | 24 weeks
  Transient elastography
Change in waist circumference | 24 weeks
Change in body weight | 24 weeks
Systolic blood pressure | 24 weeks
Diastolic blood pressure | 24 weeks
Mean arterial pressure | 24 weeks
Percentage of extracellular fluid | 24 weeks
  Bioimpedance analysis

OTHER OUTCOMES:
Change in kidney oxygenation (R2*) | 24 weeks
  Assessed via blood oxygenation dependent magnetic resonance imaging (BOLD-MRI) in an optional cohort.
Change in kidney fibrosis (ADC) | 24 weeks
  Assessed via blood oxygenation dependent magnetic resonance imaging (BOLD-MRI) in an optional cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Singh, MD MSc FRCPC, Principal Investigator — University Health Network, Toronto General Hospital
Locations (2):
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No